CLINICAL TRIAL: NCT07340437
Title: Clinical Study of an ¹⁸F-labeled GLP-1R Probe in Insulinoma
Brief Title: Clinical Study of 18F-Exendin-4 in Insulinoma
Status: Completed | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Principal Investigator, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPH-Insulinoma
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Insulinoma
MeSH Terms: conditions — Insulinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the diagnostic value of ¹⁸F-Exendin-4 PET/CT imaging in renal insulinoma. Participants will undergo clinical evaluation and ¹⁸F-Exendin-4 PET/CT examination.

DETAILED DESCRIPTION:
Early detection, precise diagnosis, and accurate localization are key to the effective management of insulinoma, the most common functional pancreatic neuroendocrine tumor, which is predominantly benign. Histopathological examination remains the diagnostic gold standard, but invasive procedures such as biopsy carry risks of bleeding and hematoma, while rarer complications like infection or pancreatic fistula may also occur. Therefore, there is an urgent clinical need for a highly accurate, non-invasive diagnostic method.

The glucagon-like peptide-1 receptor is overexpressed in insulinomas, making GLP-1R-targeted imaging a major focus in the molecular imaging of this disease. Exendin-4, an analog of GLP-1R agonists, has been shown to specifically bind to GLP-1R when labeled with ⁶⁸Ga, enabling targeted diagnosis of insulinoma. However, compared to ⁶⁸Ga, ¹⁸F offers significant advantages. Although ¹⁸F-labeled exendin-4 has been explored in preclinical studies, its clinical translation has not yet been reported. Therefore, investigating the imaging performance of ¹⁸F-exendin-4 PET/CT in insulinoma is of high clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* biochemically confirmed hyperinsulinemic hypoglycemia (plasma glucose < 3.0 mmol/L, insulin > 3 μIU/mL, C-peptide > 0.6 ng/mL)
* surgical or biopsy-confirmed insulinoma or non-insulinoma pancreatogenous hypoglycemia syndrome, with definitive clinical diagnosis at discharge and comprehensive evaluation for hypoglycemia etiology during hospitalization.

Exclusion Criteria:

* unknown etiology of hypoglycemia at last follow-up
* patients clinically diagnosed with insulinoma but without subsequent surgical intervention or biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed or highly suspected insulinoma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between clinical indicators and PET/CT results | 2 years
  Correlation analysis of clinical biochemical indicators, endoscopic ultrasound, contrast-enhanced CT, contrast-enhanced MRI with ¹⁸F-Exendin-4 PET/CT results.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Department of Nuclear Medicine, Sichuan Provincial People's Hospital, Chengdu, Sichuan 610072, Chengdu, China